CLINICAL TRIAL: NCT07071155
Title: A Pilot Study of Momelotinib in Combination With Hypomethylating Agent for Chronic Phase Myelodysplastic Syndromes/Myeloproliferative Overlap Neoplasms and Chronic Neutrophilic Leukemia (M-HArbOr)
Brief Title: Momelotinib in Combination With Hypomethylating Agent for Chronic Phase Myelodysplastic Syndromes/Myeloproliferative Overlap Neoplasms and Chronic Neutrophilic Leukemia
Acronym: M-HArbOr
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2586; IRB00509021 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes; Myeloproliferative Overlap Neoplasms; Chronic Neutrophilic Leukemia
Keywords: momelotinib; chronic neutrophilic leukemia; myelodysplastic; myeloproliferative
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Neutrophilic, Chronic | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide; Azacitidine

STUDY DESIGN:
Intervention Model Description: This is an open-label study of MMB-HMA in MDS/MPN and CNL. The investigators will enroll a total of 18 evaluable patients using a modified 3+3 dose escalation design followed by expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination therapy (MMB-HMA) (Experimental): Combination of once daily oral momelotinib plus hypomethylating agents (HMA), e.g. azacitidine) starting cycle 1. Azacitidine will be administered as an injection at 75 mg/m2 for days 1-5 in a 28-day cycle.
  Dose escalation Phase:
  The first 3 patients will receive MMB 150 mg daily in combination with azacitidine. Depending on the number of dose limiting toxicities (DLTs) experienced during this period, participants in this phase of the study will receive either 150mg daily or have an escalated dose of 200mg daily. Depending on DLT assessment during this phase of the study, the maximum tolerated dose (MTD) of either 150mg or 200mg will be determined.
  Expansion Phase:
  Once the MTD is determined (either 150 mg or 200 mg), all remaining patients up to the total of 18 evaluable patients will be treated at the MTD.
  Interventions: Drug: Momelotinib; Drug: Azacitidine

INTERVENTIONS:
Drug: Momelotinib — Capsules of Momelotinib will be administered orally once a day by all participants for up to 24 months, depending on response to treatment.
  Dose escalation will include the first 3 patients who will receive either 150 mg or 200mg of momelotinib daily, depending on the number of dose limiting toxicities (DLTs) experienced during this period.
  Dose expansion will include up to 18 evaluable participants who will receive the maximum tolerated dose (either 150mg or 200 mg) daily as will be determined during the dose escalation phase.
  Other Names: OJJAARA
Drug: Azacitidine — 75 mg/m2, days 1-5 in a 28-day cycle
  Other Names: Vidaza

SUMMARY:
This research is being done to evaluate effectiveness, safety, and tolerability of a study drug called momelotinib in participants with myelodysplastic/myeloproliferative neoplasms (MDS/MPNs), MDS/MPN-not otherwise specified (MDS/MPN-NOS), MDS/MPN with neutrophilia (MDS/MPN-N), also called as atypical chronic myeloid leukemia, or chronic neutrophilic leukemia. Momelotinib will be added to standard treatment which usually includes a hypomethylating agent like azacitidine. Treatment options for this diagnosis remain limited and investigators need better treatments to help control the disease, improve symptoms, and potentially help more patients become eligible for transplant.

Participants for this study will be asked to take some screening tests which will include routine physical examination, blood tests, and imaging scans to determine eligibility for the study. Those who continue to qualify for this study will begin treatment and may be asked to remain on the study drug for up to 24 months, depending upon how they are responding to treatment. After the study drug is completed, patients will have one additional clinic visit to evaluate overall health and response to study drug. The study drug treatment on this study will include taking momelotinib by mouth in combination with azacitidine, which is given by injection for all patients for the first 5 days of each 28-day cycle.

The most common side effect that may be related to participation in this study can include (i) infections which can present as fever, chills, cough, breathing problems, diarrhea, vomiting, pain or burning with urination; or (ii) low blood platelet count which can result in bruising or bleeding for longer than usual if the participant hurts themself.

DETAILED DESCRIPTION:
This is an open-label study of MMB-HMA in MDS/MPN and CNL that will enroll up to 18 patients. Momelotinib will be administered using modified 3+3 dose escalation design followed by expansion. The first three patients will be treated at 150mg daily and if DLT criteria are not met, the remaining patients will be treated at 200mg daily to a total of 18 evaluable patients (all in combination with azacitidine). If DLTs are met within the dose escalation phase (first three patients), then the patients will be treated at 150mg daily (in combination with azacitidine)

Key Eligibility Criteria:

1. Patients with a WHO diagnosis of chronic myelomonocytic leukemia (CMML), MDS/MPN-not otherwise specified (MDS/MPN-NOS), MDS/MPN with neutrophilia (MDS/MPN-N), CNL.
2. Age greater than or equal to 18 years
3. Blood counts with platelets greater than 25,000/microL, ANC greater than or equal to 0.75 x 10^9/L (without transfusion or growth factor support)
4. Baseline splenomegaly with greater than or equal to 5 cm below costal margin or greater than or equal to 450 cm3 on imaging (ultrasound, CT or MRI)

ELIGIBILITY:
* Patients of age 18 or older
* Has a diagnosis of MDS/MPN or CNL by WHO or ICC diagnostic criteria:

  1. Chronic myelomonocytic leukemia
  2. MDS/MPN with neutrophilia, previously known as atypical chronic myeloid leukemia
  3. Chronic neutrophilic leukemia
  4. MDS/MPN -not otherwise specified
* Chronic phase disease with <10% blasts in peripheral blood and marrow within 1 month from planned start of treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Score44 of 0-2
* Patients can be treatment naïve or could have undergone prior treatments for MDS/MPN as below:

  1. Prior treatment with non-JAK inhibitors or hypomethylating agents are allowed (e.g., hydroxyurea, immunomodulatory agents, steroids). Hydroxyurea can be continued until or even beyond initiation of treatment for 2 months if needed for cytoreduction
  2. If non-MMB JAK inhibitors were used for treatment and stopped due to side effects (e.g., anemia from ruxolitinib, gastrointestinal toxicity from fedratinib, etcetera), these patients will be allowed to enroll on this study as long as JAK inhibitor was stopped at least 2 weeks prior to anticipated start date of treatment
  3. If prior hypomethylating agent was used and stopped longer than 3 months prior to anticipated start date of treatment due to side effects, these patients will be eligible. However, if hypomethylating agents were stopped due to lack of clinical benefit, these patients will not be deemed eligible
  4. Prior treatment with erythropoietic stimulating agents is allowed if last treatment was more than 4 weeks prior to anticipated start date of treatment
  5. Splenic radiation should have been performed more than 2 months before anticipated start date of treatment
  6. Any prior or ongoing investigation therapy or agents should be stopped longer than 4 weeks of anticipated start date of treatment
* Blood counts with platelets ≥25,000/microL, ANC ≥0.75 x 10^9/L (without transfusion or growth factor support)
* Baseline splenomegaly with ≥5 cm below costal margin or ≥450 cm3 on imaging (ultrasound, CT or MRI)
* Adequate organ function with creatinine clearance measured by Cockcroft-Gault calculation ≥30 mL/min, total bilirubin ≤1.5×ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%), INR ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within the therapeutic range of intended use of anticoagulants, albumin ≥2.5 g/dL.
* Willing and able to sign the informed consent form
* Life expectancy > 24 weeks
* Willing and able to complete patient-reported outcome assessments using an ePRO device according to protocol
* Patients of child-bearing potential, or those with partners of child-bearing potential or pregnant or lactating partners, who are willing to follow highly effective contraceptive requirements. Females of reproductive potential should use effective contraception during study treatment and for 6 months following the last dose for HMA-MMB and 1 week following the last dose for MMB monotherapy. Males with female partners of reproductive potential should use effective contraception during study treatment and for 3 months following the last dose for HMA-MMB and 1 week following the last dose for MMB monotherapy. Patients should not breastfeed during treatment and for 1 week after the last dose.
* Patients of child-bearing potential with a negative highly sensitive serum pregnancy test within 24 hours before the first dose of momelotinib.

Exclusion criteria

* Diagnosis of MDS/MPN with SF3B1 gene mutation and thrombocytosis (excluded due to unclear role of ACRV1 in the development of anemia)
* Peripheral blood or marrow (by immunohistochemistry) blast percentage >10%
* Prior lack of response to MMB or hypomethylating agents.
* Known history of allergic reaction to momelotinib
* AST or ALT above 2.5 x ULN (above 5 X ULN if liver is involved by extramedullary hematopoiesis as judged by the investigator or if related to iron chelator therapy that was started within the prior 60 days)
* The following treatments within the time periods as specified:

  1. Momelotinib at any time prior to screening
  2. Erythropoietic stimulating agents within 4 weeks of treatment
  3. Investigational agent within 4 weeks of the first dose of study treatment
  4. Immunosuppressive agents within 28 days (low dose steroids ≤10 mg daily prednisone or equivalent is allowed)
  5. Potent cytochrome P450 3A4 (CYP3A4) inducers, except for rifampin and rifampicin, within 14 days prior to the first dose of momelotinib. Strong CYP3A4 inducers can lead to decreased MMB exposure and risk a lack of efficacy. Therefore, alternative medicinal product to strong CYP3A4 inducer should be considered.
* Unsuitable for spleen volume measurements due to prior splenectomy or unwilling or unable to undergo any imaging (ultrasound, CT without contrast or MRI without contrast) for spleen volume measurement per requirements
* Patients with an active invasive concurrent malignancy, whose natural history or treatment has a significant potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Localized prostate cancer that has been treated surgically or by radiotherapy with curative intent and presumed cured is allowed.
* History of non-melanoma skin cancers such as basal cell carcinoma or squamous cell carcinoma are also allowed.
* Completely resected intraepithelial carcinoma of cervix or papillary thyroid or follicular thyroid cancers are also allowed at the investigator's discretion.
* Untreated or active infections are excluded as below:

  1. Chronic active or acute viral hepatitis A, B, or C infection. Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative hepatitis C RNA test is obtained.
  2. HIV with CD4+ cell count under 400 cells/ μL or on treatment with anti-retroviral therapy that is specifically excluded per the criteria above. HIV patients on established anti-retroviral therapy allowed per protocol for at least 4 weeks and CD4+ count above or equal to 400 cells/ μL
  3. Infections requiring intravenous antibiotics
* Nonhematologic toxicities from prior therapies that are unresolved and are of grade >1
* Presence of peripheral neuropathy of grade ≥2
* Pregnant women are excluded from this study because the effects of momelotinib on embryotoxicity, survival, and teratogenicity remain unclear.
* Patients unable to swallow medications
* Patient has any medical condition that puts the patient at an acceptable high risk with participation in the study per physician assessment or has any condition that confounds the ability to interpret data from the study.
* Any major surgery or radiation or intervention that interferes with safety or feasibility of enrollment per investigator assessment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-03-05 (Estimated); Primary Completion 2028-03-05 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve a complete response | 24 weeks
  Efficacy determination - complete response: number of participants who achieve a complete response as defined by international consortium response criteria for MDS/MPN in adults
Number of participants who achieve a partial response | 24 weeks
  Efficacy determination - partial response: number of participants who achieve a partial response as defined by international consortium response criteria for MDS/MPN in adults
Number of participants who achieve a clinical benefit | 24 weeks
  Efficacy determination - clinical benefit: number of participants who achieve a clinical benefit per MDS/MPN IWG criteria4

SECONDARY OUTCOMES:
Number of participants who experience a grade 3 or higher adverse events or severe event | 2 years
  Safety and tolerability evaluation: number of participants who experience a grade 3 or higher adverse event events or severe adverse events as defined by CTCAE v.5.0
Number of Participants Who Achieve Erythroid Response | 12 weeks
  Number of patients who achieve erythroid response at week 12 per international consortium criteria
Number of Participants Who Achieve Erythroid Response | 24 weeks
  Number of participants who achieve erythroid response at week 24 per international consortium criteria
Proportion of Participants Who Achieve Spleen Size Reduction | 12 weeks
  Determine the proportion of participants who achieve a spleen volume reduction of ≥ 35% from baseline at week 12
Proportion of participants Who Achieve Spleen Size Reduction | 24 weeks
  Determine the proportion of participants who achieve a spleen volume reduction of ≥ 35% from baseline at week 24
Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) | 12 weeks
  Evaluate efficacy of momelotinib plus hypomethylating agents azacitidine or decitabine (MMB-HMA) on MPN-SAF TSS questionnaire. Score range 0-100, higher score worse symptoms.
Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) | 24 weeks
  Evaluate efficacy of momelotinib plus hypomethylating agents azacitidine or decitabine (MMB-HMA) on MPN-SAF TSS questionnaire. Score range 0-100, higher score worse symptoms.
Patient Global Impression of Change (PGIC) questionnaire | 12 weeks
  Evaluate efficacy of momelotinib plus hypomethylating agents azacitidine or decitabine (MMB-HMA) on Patient Global Impression of Change (PGIC) questionnaire. A 7-point scale (1-7) rating of overall improvement. Patients rate their change as 1="very much improved," 2="much improved," 3="minimally improved," 4="no change," 5="minimally worse," 6="much worse," or 7="very much worse." Lower values represent a better outcome.
Patient Global Impression of Change (PGIC) | 24 weeks
  Evaluate efficacy of momelotinib plus hypomethylating agents azacitidine or decitabine (MMB-HMA) on Patient Global Impression of Change (PGIC) questionnaire. A 7-point scale (1-7) rating of overall improvement. Patients rate their change as 1="very much improved," 2="much improved," 3="minimally improved," 4="no change," 5="minimally worse," 6="much worse," or 7="very much worse." Lower values represent a better outcome.
Trough concentrations of MMB as single agent and in combination with HMA | 12 weeks
  Evaluate trough concentrations at week 12 in Arm A and B
Trough concentrations of MMB as single agent and in combination with HMA | 24 weeks
  Evaluate trough concentrations at week 24 in Arm A and B

CONTACTS AND LOCATIONS:
Overall Officials: Tania Jain, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT07071155/Prot_SAP_000.pdf